CLINICAL TRIAL: NCT04864041
Title: Evaluation of Left Ventricular Function by Speckle Tracking Echocardiography in Patient Hospitalised in Intensive Care Unit for Vaso-occlusive Crisis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Clinical Professor, Bicetre Hospital
Other Study IDs: 2021-A00623-38
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Sickle Cell Disease
Keywords: ICU Intensive Care Units; Transthoracic Echocardiography; Left Ventricular Function
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalised in ICU for vaso-occlusive crisis
  Interventions: Other: Evaluation of global longitudinal strain using routinely recorded echocardiography images

INTERVENTIONS:
Other: Evaluation of global longitudinal strain using routinely recorded echocardiography images — There are no particular intervention performed in patients in this study, because echocardiography is part of the standard of care of patients hospitalised in the ICU for vaso occlusive crisis.

SUMMARY:
Vaso-occlusive crisis in Sickle cell disease might alter myocardial function through micro vascular obstruction. Evaluation of strain alteration using speckle tracking echocardiography is a non invasive technique that may allow us to observe such myocardial dysfunction. No such study has yet been conducted in patient hospitalised in intensive care unit. Our hypothesis is that strain alteration during vaso-occlusive crisis, if they do exist, can be correlated with other markers of myocardial injury such as troponin level or thoracic pain.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation in an intensive care unit for vaso-occlusive crisis

Exclusion Criteria:

* Pregnancy
* Individuals under guardianship
* Unsufficient echogenicity
* Thoracic pain prohibiting echocardiography assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with vaso occlusive crisis hospitalised in an intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Global longitudinal strain | Day 0
  Measure of global longitudinal strain using speckle tracking echocardiography
Global longitudinal strain | Day 1
  Measure of global longitudinal strain using speckle tracking echocardiography
Global longitudinal strain | Day 2
  Measure of global longitudinal strain using speckle tracking echocardiography

SECONDARY OUTCOMES:
Troponine level | Day 0
Troponine level | Day 1
Troponine level | Day 2
Electrocardiogram QT interval | Day 0
Electrocardiogram QT interval | Day 2
Electrocardiogram ST elevation | Day 0
Electrocardiogram ST elevation | Day 2
Electrocardiogram negative T waves | Day 0
Electrocardiogram negative T waves | Day 2
Thoracic pain | Day 0
  Numerical rating scale from 0 to 10 assessed by the patient
Thoracic pain | Day 1
  Numerical rating scale from 0 to 10 assessed by the patient
Thoracic pain | Day 2
  Numerical rating scale from 0 to 10 assessed by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No